CLINICAL TRIAL: NCT05765786
Title: Do we Miss a Common Subset of Primary Aldosteronism in Which There is Cyclical or Exaggerated Diurnal Variation in Secretion?
Brief Title: Diagnosing Variable Primary Aldosteronism.
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 318689
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Primary Aldosteronism; High Blood Pressure
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and whole blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to see if there is a cyclical or exaggerated diurnal variation in aldosterone production in people with Primary Aldosteronism.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

* Can we diagnose more people if we used 24 hour urine measurements?
* In those with high amounts of aldosterone in their urine, is there a variable pattern to their aldosterone production?

Participants will have a 24 hour urine measurement. They will also have multiple blood tests throughout the day to study the variability in aldosterone secretion.

ELIGIBILITY:
Inclusion Criteria:

* People with clinically suspected PA but have not met criteria for diagnosis. Suspicion based on low-renin (renin activity <0.5 nmol/h/L or renin mass <5 ng/L), plasma sodium > 140mmol/L or plasma potassium < 4mmol/L.
* Patients who have been diagnosed with PA and had previous aldosterone samples <277 pmol/L, a level which would normally not qualify for confirmatory testing.
* Patients with aldosterone results done at different times that indicate variability in production.
* Willing to consent and participate in the study.

Exclusion Criteria:

* Inability to withdraw β-adrenoceptor antagonist therapy for 2 weeks.
* People on end of life treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 24 hour urine tetrahydroaldosterone excretion. | 12 months
  Can measurement of 24 hour urine tetrahydroaldosterone excretion detect more people with PA than current conventional screening tests?

SECONDARY OUTCOMES:
Differences in timed day and night urine THA measurements. | 12 months
  We will be measuring the 24 hour urine THA samples in two separate (approximately 12 hours each) collections, one in the day and one at night. We can then study if there are any differences between day time and night time secretion which may help us understand the diurnal variation in aldosterone secretion.
Variation in aldosterone secretion from day series in those with positive 24h urine THA and those with negative 24h urine THA. | 12 months
  This will allow us to study further if the reason why their screening blood test did not meet the threshold for diagnosis.
Complete or partial clinical cure rate of this cohort of patients that qualify for adrenalectomy | 12 months
  Complete clinical cure is daytime home or ambulatory BP < 135/<85mmHg, on no treatment. Partial clinical cure is BP < 135/<85 mmHg on the same or fewer drugs, not including a K+-sparing diuretic.
Complete biochemical cure of PA in this cohort of patients that qualify for adrenalectomy. | 12 months
  This is defined as (whilst off medications that might alter serum potassium or the RAS) by both:
  1. normalization of serum potassium and normalization of ARR or
  2. elevated ARR and either baseline PAC <190pmol/L, or normal confirmatory test (saline infusion test or captopril challenge test).

CONTACTS AND LOCATIONS:
Overall Officials: William Drake, Prof, Principal Investigator — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom